CLINICAL TRIAL: NCT02384395
Title: IGHID 11417 - The Safety and Efficacy of Fixed Dose Combination Dolutegravir/Abacavir/Lamivudine FDC Initiated During Acute HIV Infection: Impact on the Latent HIV Reservoir and Long-Term Immunologic Effect
Brief Title: Safety and Efficacy of Fixed Dose Combination Dolutegravir/Abacavir/Lamivudine FDC Initiated During Acute HIV Infection
Acronym: PHI-05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-0549
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: HIV; Acute HIV Infection
Keywords: Dolutegravir; Abacavir; Lamivudine; acute HIV infection; human leukocyte antigen; latent HIV reservoir; integrase-based regimen; viremia; antiretroviral therapy; fixed dose combination
MeSH Terms: conditions — Viremia | interventions — dolutegravir; Lamivudine; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DTG/3TC/ABC FDC (Experimental): Dolutegravir (DTG 50 mg), abacavir sulfate (ABC 600 mg) and lamivudine (3TC 300 mg) formulated in a single tablet fixed dose combination (FDC) (DTG/ABC/3TC, GSK2619619), administered orally, once daily
  Interventions: Drug: Dolutegravir 50 mg; Drug: Lamivudine 300 mg; Drug: Abacavir 600 mg

INTERVENTIONS:
Drug: Dolutegravir 50 mg — Initial therapy for AHI
  Other Names: DTG; Tivicay
Drug: Lamivudine 300 mg — Initial therapy for AHI
  Other Names: 3TC; Epivir
Drug: Abacavir 600 mg — Initial therapy for AHI
  Other Names: ABC; Ziagen

SUMMARY:
This is a multicenter, single arm, 96-week open-label study of the safety and virologic efficacy of fixed dose combination Dolutegravir/Lamivudine/Abacavir (DTG/3TC/ABC FDC) initiated during acute HIV infection (AHI).

DETAILED DESCRIPTION:
The study will be conducted at the University of North Carolina in Chapel Hill, NC and Duke University in Durham, NC. The investigators plan to enroll up to 44 participants who will be enrolled for 96 weeks and will receive DTG/3TC/ABC FDC.

The investigators propose to evaluate the efficacy and time to viral suppression with DTG/3TC/ABC FDC as initial therapy for acute HIV infection (AHI), as well as the feasibility of prompt administration using a rapid human leukocyte antigen-B57 (HLA-B57) screening antibody assay. In addition to validating the restriction of resting cell infection (RCI) by antiretroviral therapy (ART) including a DTG-based regimen initiated during AHI, the investigators will seek correlations between low RCI, residual gastrointestinal associated lymphoid tissue (GALT) HIV expression, and measures of immune activation. The investigators hypothesize that rapid reduction in plasma viremia with this regimen will limit the area under the pre-ART viral load curve, and thus reduce the latent reservoir size as measured by a viral outgrowth assay one to two years following ART start, and as compared with the latent reservoir size in acutely infected individuals started on regimens without an integrase inhibitor based regimen. In addition, the investigators will examine the longitudinal impact of the proposed integrase-based regimen initiated during the acute period on immune activation through week 96. If residual viral expression and persistent immune dysfunction is related to the burden of the latent viral reservoir (and presumably its periodic activation) these abnormalities should be ameliorated by early ART with rapid viral suppression. The investigators hypothesize that earlier treatment coupled with more rapid ART-mediated virus suppression will be associated with better long-term T cell function, specifically better T cell function after 2 years of durable HIV suppression.

ELIGIBILITY:
Inclusion Criteria

1. Documentation of Acute HIV infection at or within 30 days of study entry.
2. Men and women age ≥18 years.
3. ART naive, defined as ≤14 days of antiretroviral treatment at any time prior to entry. The only exceptions are:

   * Pre-exposure prophylaxis (PrEP) and documented as HIV-1 negative at least 1 month prior to AHI diagnosis during PrEP, and
   * Post-exposure prophylaxis (PEP) provided the participant was documented as HIV-1 negative at least 3-6 months following completion of PEP treatment.
4. Lab values obtained within 30 days prior to study entry:

   * Absolute neutrophil count >500/mm^3
   * Hemoglobin > 8.5 g/dL for men and > 8.0 g/dL for women
   * Platelet count >50,000/mm^3
   * Lipase ≤ 3 X upper limit of normal (ULN), single repeat test is allowed to determine eligibility
   * Calculated creatinine clearance (CrCl, Cockcroft-Gault formula) ≥ 50 mL/min:

   CrCl = (140-age) x body weight (kg) (x 0.85 if female) Serum creatinine [mg/dL] x (72)
5. Testing for HBsAg is pending. Note: Participants who test positive for HBsAg will be terminated from the study prior to starting study treatment.
6. Testing for HLA-B57 and/or HLA-B*5701 is pending. Note: Participants who test positive for HLA-B*5701 will be terminated from the study prior to starting study treatment.
7. A female is eligible to enter and participate in the study if she:

   * Is of non-childbearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy; or,
   * Is of child-bearing potential, with a negative pregnancy test at screening and at enrollment, who agrees to use one of the methods of contraception listed below.
   * Complete abstinence from intercourse from 2 weeks prior to administration of study medication, throughout the study, and for at least 2 weeks after discontinuation of all study medication;
   * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
   * Approved hormonal contraception - used alone is not considered a sufficient form of contraception for the study see Protocol Appendix 1 for a listing of examples of approved hormonal contraception;
   * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year; see Protocol Appendix 2 for a listing of IUDs meeting this criterion;
   * Male partner sterilization confirmed prior to the female participant's entry into the study, and this male is the sole partner for that patient;
   * Any other method with published data showing that the expected failure rate is <1% per year.
   * Any contraception method must be used consistently, in accordance with the approved product label and for at least 2 weeks after discontinuation of the study medication.
8. Females who meet the post-menopausal definition, noted in inclusion criterion 7, will have a follicle stimulation hormone (FSH) test to verify menopause,
9. Ability and willingness of participant to give written informed consent.

Exclusion Criteria

1. Alanine Transaminase (ALT) ≥ 5 times Upper Limit of Normal (≥5xULN)
2. Aspartate Aminotransferase (AST) ≥ 3x ULN
3. Bilirubin ≥1.5x ULN (with >35% direct bilirubin)
4. Weight <40 kg
5. Women who are breast-feeding.
6. Women with a positive pregnancy test on enrollment or prior to study drug administration.
7. Women and men of child bearing potential unwilling to agree to use an effective methods of contraception required by the study.
8. History or presence of allergy to the study drugs or their components.
9. Requires or is anticipated to require any of the prohibited concomitant therapy: barbiturates, dofetilide, fampridine (dalfampridine), modafinil, oxcarbazepine, pioglitazone, pilsicainide, pimozide, rifampin, rifapentine, phenytoin, phenobarbital, carbamazepine, and St. John's wort.

   * Dofetilide, fampridine, and pilsicainide are prohibited, as DTG may inhibit its renal tubular secretion resulting in increased dofetilide concentrations and potential for toxicity.
10. Unable to discontinue any current medications that are excluded during study treatment.
11. Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), radiation therapy, HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry.

    * Prednisone at a daily dose of 10 mg or less (physiologic replacement dose) is permitted.
12. Treatment with radiation therapy or cytotoxic chemotherapeutics agents within 28 days prior to screening or has an anticipated need for these agents during the study.
13. Administration of an HIV-1 immunotherapeutic vaccine within 90 days prior to screening.
14. Prior treatment with any other experimental drug for any indication (within 30 days of initiating study treatment).
15. Difficulty swallowing capsules/tablets.
16. Inability to communicate effectively with study personnel.
17. Incarceration; prisoner recruitment and participation are not permitted.
18. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements or confound the analysis of study endpoints.
19. Any condition (including but not limited to alcohol and drug use) or any active clinically significant disease or findings during screening of medical history or physical examination, which, in the opinion of the Investigator would interfere with patient safety or compliance.
20. Serious illness requiring systemic treatment and/or hospitalization until patient either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry.

    Note: Oral candidiasis, vaginal candidiasis, mucocutaneous herpes simplex, and other minor illnesses (as judged by the site investigator) have no restriction.
21. A life expectancy less than twelve months.
22. Acute viral hepatitis, including, but not limited to, hepatitis A, B, or C.
23. History of myocardial infarction or diagnosis of coronary artery disease.
24. History of ongoing or clinically relevant pancreatitis within the previous 6 months.
25. Chronic hepatitis C infection with an anticipated need for treatment during the study period (through week 96).
26. Chronic hepatitis B infection (see inclusion criterion 5).
27. Evidence for moderate to severe hepatic impairment (as defined by the presence of cirrhosis, ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice or Child-Pugh class B or greater hepatic impairment).
28. Evidence of biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
29. Any verified grade 4 laboratory abnormality with exception of ALT as defined in exclusion criterion 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2020-03-06 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Gay, MD, MPH, Principal Investigator — University of North Carolina
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adolescents. PoAGfAa. Guidelines for the use of antiretroviral agents in HIV-1-infected adults and adolescents. In: Department of Health and Human Servies.; 2013
- [Background] Ortiz GM, Nixon DF, Trkola A, Binley J, Jin X, Bonhoeffer S, Kuebler PJ, Donahoe SM, Demoitie MA, Kakimoto WM, Ketas T, Clas B, Heymann JJ, Zhang L, Cao Y, Hurley A, Moore JP, Ho DD, Markowitz M. HIV-1-specific immune responses in subjects who temporarily contain virus replication after discontinuation of highly active antiretroviral therapy. J Clin Invest. 1999 Sep;104(6):R13-8. doi: 10.1172/JCI7371. PMID 10491418
- [Background] Pilcher CD, Eron JJ Jr, Galvin S, Gay C, Cohen MS. Acute HIV revisited: new opportunities for treatment and prevention. J Clin Invest. 2004 Apr;113(7):937-45. doi: 10.1172/JCI21540. PMID 15057296
- [Background] Pires A, Hardy G, Gazzard B, Gotch F, Imami N. Initiation of antiretroviral therapy during recent HIV-1 infection results in lower residual viral reservoirs. J Acquir Immune Defic Syndr. 2004 Jul 1;36(3):783-90. doi: 10.1097/00126334-200407010-00004. PMID 15213561
- [Background] Ramratnam B, Ribeiro R, He T, Chung C, Simon V, Vanderhoeven J, Hurley A, Zhang L, Perelson AS, Ho DD, Markowitz M. Intensification of antiretroviral therapy accelerates the decay of the HIV-1 latent reservoir and decreases, but does not eliminate, ongoing virus replication. J Acquir Immune Defic Syndr. 2004 Jan 1;35(1):33-7. doi: 10.1097/00126334-200401010-00004. PMID 14707789
- [Background] Chamberland A, Sylla M, Boulassel MR, Baril JG, Cote P, Thomas R, Trottier B, Rouleau D, Routy JP, Tremblay C; Investigators of the Primary HIV-Infection Cohort of Montreal. Effect of antiretroviral therapy on HIV-1 genetic evolution during acute infection. Int J STD AIDS. 2011 Mar;22(3):146-50. doi: 10.1258/ijsa.2010.010292. PMID 21464451
- [Background] Gay CL, Mayo AJ, Mfalila CK, Chu H, Barry AC, Kuruc JD, McGee KS, Kerkau M, Sebastian J, Fiscus SA, Margolis DM, Hicks CB, Ferrari G, Eron JJ; Duke-UNC Acute HIV Infection Consortium. Efficacy of NNRTI-based antiretroviral therapy initiated during acute HIV infection. AIDS. 2011 Apr 24;25(7):941-9. doi: 10.1097/QAD.0b013e3283463c07. PMID 21487250
- [Background] Cossarini F, Boeri E, Canducci F, Salpietro S, Bigoloni A, Galli L, Spagnuolo V, Castagna A, Clementi M, Lazzarin A, Gianotti N. Integrase and fusion inhibitors transmitted drug resistance in naive patients with recent diagnosis of HIV-1 infection. J Acquir Immune Defic Syndr. 2011 Feb 1;56(2):e51-4. doi: 10.1097/QAI.0b013e3181fcc0f1. No abstract available. PMID 21233631
- [Background] Markowitz M, Nguyen BY, Gotuzzo E, Mendo F, Ratanasuwan W, Kovacs C, Prada G, Morales-Ramirez JO, Crumpacker CS, Isaacs RD, Campbell H, Strohmaier KM, Wan H, Danovich RM, Teppler H; Protocol 004 Part II Study Team. Sustained antiretroviral effect of raltegravir after 96 weeks of combination therapy in treatment-naive patients with HIV-1 infection. J Acquir Immune Defic Syndr. 2009 Nov 1;52(3):350-6. doi: 10.1097/QAI.0b013e3181b064b0. PMID 19648823
- [Background] Cohen C, Elion R, Ruane P, Shamblaw D, DeJesus E, Rashbaum B, Chuck SL, Yale K, Liu HC, Warren DR, Ramanathan S, Kearney BP. Randomized, phase 2 evaluation of two single-tablet regimens elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate versus efavirenz/emtricitabine/tenofovir disoproxil fumarate for the initial treatment of HIV infection. AIDS. 2011 Mar 27;25(6):F7-12. doi: 10.1097/QAD.0b013e328345766f. PMID 21412057
- [Background] Archin NM, Vaidya NK, Kuruc JD, Liberty AL, Wiegand A, Kearney MF, Cohen MS, Coffin JM, Bosch RJ, Gay CL, Eron JJ, Margolis DM, Perelson AS. Immediate antiviral therapy appears to restrict resting CD4+ cell HIV-1 infection without accelerating the decay of latent infection. Proc Natl Acad Sci U S A. 2012 Jun 12;109(24):9523-8. doi: 10.1073/pnas.1120248109. Epub 2012 May 29. PMID 22645358
- [Background] Vinikoor MJ, Cope A, Gay CL, Ferrari G, McGee KS, Kuruc JD, Lennox JL, Margolis DM, Hicks CB, Eron JJ. Antiretroviral therapy initiated during acute HIV infection fails to prevent persistent T-cell activation. J Acquir Immune Defic Syndr. 2013 Apr 15;62(5):505-8. doi: 10.1097/QAI.0b013e318285cd33. PMID 23314410
- [Background] Lennox JL, Dejesus E, Berger DS, Lazzarin A, Pollard RB, Ramalho Madruga JV, Zhao J, Wan H, Gilbert CL, Teppler H, Rodgers AJ, Barnard RJ, Miller MD, Dinubile MJ, Nguyen BY, Leavitt R, Sklar P; STARTMRK Investigators. Raltegravir versus Efavirenz regimens in treatment-naive HIV-1-infected patients: 96-week efficacy, durability, subgroup, safety, and metabolic analyses. J Acquir Immune Defic Syndr. 2010 Sep;55(1):39-48. doi: 10.1097/QAI.0b013e3181da1287. PMID 20404738
- [Background] Raffi F, Rachlis A, Stellbrink HJ, Hardy WD, Torti C, Orkin C, Bloch M, Podzamczer D, Pokrovsky V, Pulido F, Almond S, Margolis D, Brennan C, Min S; SPRING-2 Study Group. Once-daily dolutegravir versus raltegravir in antiretroviral-naive adults with HIV-1 infection: 48 week results from the randomised, double-blind, non-inferiority SPRING-2 study. Lancet. 2013 Mar 2;381(9868):735-43. doi: 10.1016/S0140-6736(12)61853-4. Epub 2013 Jan 8. PMID 23306000
- [Background] Siliciano JD, Kajdas J, Finzi D, Quinn TC, Chadwick K, Margolick JB, Kovacs C, Gange SJ, Siliciano RF. Long-term follow-up studies confirm the stability of the latent reservoir for HIV-1 in resting CD4+ T cells. Nat Med. 2003 Jun;9(6):727-8. doi: 10.1038/nm880. Epub 2003 May 18. PMID 12754504
- [Background] Archin NM, Eron JJ, Palmer S, Hartmann-Duff A, Martinson JA, Wiegand A, Bandarenko N, Schmitz JL, Bosch RJ, Landay AL, Coffin JM, Margolis DM. Valproic acid without intensified antiviral therapy has limited impact on persistent HIV infection of resting CD4+ T cells. AIDS. 2008 Jun 19;22(10):1131-5. doi: 10.1097/QAD.0b013e3282fd6df4. PMID 18525258
- [Background] Archin NM, Cheema M, Parker D, Wiegand A, Bosch RJ, Coffin JM, Eron J, Cohen M, Margolis DM. Antiretroviral intensification and valproic acid lack sustained effect on residual HIV-1 viremia or resting CD4+ cell infection. PLoS One. 2010 Feb 23;5(2):e9390. doi: 10.1371/journal.pone.0009390. PMID 20186346
- [Background] Chun TW, Justement JS, Moir S, Hallahan CW, Maenza J, Mullins JI, Collier AC, Corey L, Fauci AS. Decay of the HIV reservoir in patients receiving antiretroviral therapy for extended periods: implications for eradication of virus. J Infect Dis. 2007 Jun 15;195(12):1762-4. doi: 10.1086/518250. Epub 2007 May 2. PMID 17492591
- [Background] Chun TW, Stuyver L, Mizell SB, Ehler LA, Mican JA, Baseler M, Lloyd AL, Nowak MA, Fauci AS. Presence of an inducible HIV-1 latent reservoir during highly active antiretroviral therapy. Proc Natl Acad Sci U S A. 1997 Nov 25;94(24):13193-7. doi: 10.1073/pnas.94.24.13193. PMID 9371822
- [Background] Chun TW, Carruth L, Finzi D, Shen X, DiGiuseppe JA, Taylor H, Hermankova M, Chadwick K, Margolick J, Quinn TC, Kuo YH, Brookmeyer R, Zeiger MA, Barditch-Crovo P, Siliciano RF. Quantification of latent tissue reservoirs and total body viral load in HIV-1 infection. Nature. 1997 May 8;387(6629):183-8. doi: 10.1038/387183a0. PMID 9144289
- [Background] Myers LE, McQuay LJ, Hollinger FB. Dilution assay statistics. J Clin Microbiol. 1994 Mar;32(3):732-9. doi: 10.1128/jcm.32.3.732-739.1994. PMID 8195386
- [Background] Lehrman G, Hogue IB, Palmer S, Jennings C, Spina CA, Wiegand A, Landay AL, Coombs RW, Richman DD, Mellors JW, Coffin JM, Bosch RJ, Margolis DM. Depletion of latent HIV-1 infection in vivo: a proof-of-concept study. Lancet. 2005 Aug 13-19;366(9485):549-55. doi: 10.1016/S0140-6736(05)67098-5. PMID 16099290
- [Background] Koelsch KK, Boesecke C, McBride K, Gelgor L, Fahey P, Natarajan V, Baker D, Bloch M, Murray JM, Zaunders J, Emery S, Cooper DA, Kelleher AD; PINT study team. Impact of treatment with raltegravir during primary or chronic HIV infection on RNA decay characteristics and the HIV viral reservoir. AIDS. 2011 Nov 13;25(17):2069-78. doi: 10.1097/QAD.0b013e32834b9658. PMID 21860347
- [Background] Mehandru S, Poles MA, Tenner-Racz K, Jean-Pierre P, Manuelli V, Lopez P, Shet A, Low A, Mohri H, Boden D, Racz P, Markowitz M. Lack of mucosal immune reconstitution during prolonged treatment of acute and early HIV-1 infection. PLoS Med. 2006 Dec;3(12):e484. doi: 10.1371/journal.pmed.0030484. PMID 17147468
- [Background] Poles MA, Boscardin WJ, Elliott J, Taing P, Fuerst MM, McGowan I, Brown S, Anton PA. Lack of decay of HIV-1 in gut-associated lymphoid tissue reservoirs in maximally suppressed individuals. J Acquir Immune Defic Syndr. 2006 Sep;43(1):65-8. doi: 10.1097/01.qai.0000230524.71717.14. PMID 16936559
- [Background] Sax PE, DeJesus E, Mills A, Zolopa A, Cohen C, Wohl D, Gallant JE, Liu HC, Zhong L, Yale K, White K, Kearney BP, Szwarcberg J, Quirk E, Cheng AK; GS-US-236-0102 study team. Co-formulated elvitegravir, cobicistat, emtricitabine, and tenofovir versus co-formulated efavirenz, emtricitabine, and tenofovir for initial treatment of HIV-1 infection: a randomised, double-blind, phase 3 trial, analysis of results after 48 weeks. Lancet. 2012 Jun 30;379(9835):2439-2448. doi: 10.1016/S0140-6736(12)60917-9. PMID 22748591
- [Background] Steigbigel RT, Cooper DA, Kumar PN, Eron JE, Schechter M, Markowitz M, Loutfy MR, Lennox JL, Gatell JM, Rockstroh JK, Katlama C, Yeni P, Lazzarin A, Clotet B, Zhao J, Chen J, Ryan DM, Rhodes RR, Killar JA, Gilde LR, Strohmaier KM, Meibohm AR, Miller MD, Hazuda DJ, Nessly ML, DiNubile MJ, Isaacs RD, Nguyen BY, Teppler H; BENCHMRK Study Teams. Raltegravir with optimized background therapy for resistant HIV-1 infection. N Engl J Med. 2008 Jul 24;359(4):339-54. doi: 10.1056/NEJMoa0708975. PMID 18650512
- [Background] Molina JM, Lamarca A, Andrade-Villanueva J, Clotet B, Clumeck N, Liu YP, Zhong L, Margot N, Cheng AK, Chuck SL; Study 145 Team. Efficacy and safety of once daily elvitegravir versus twice daily raltegravir in treatment-experienced patients with HIV-1 receiving a ritonavir-boosted protease inhibitor: randomised, double-blind, phase 3, non-inferiority study. Lancet Infect Dis. 2012 Jan;12(1):27-35. doi: 10.1016/S1473-3099(11)70249-3. Epub 2011 Oct 18. PMID 22015077
- [Background] Rockstroh JK, DeJesus E, Lennox JL, Yazdanpanah Y, Saag MS, Wan H, Rodgers AJ, Walker ML, Miller M, DiNubile MJ, Nguyen BY, Teppler H, Leavitt R, Sklar P; STARTMRK Investigators. Durable efficacy and safety of raltegravir versus efavirenz when combined with tenofovir/emtricitabine in treatment-naive HIV-1-infected patients: final 5-year results from STARTMRK. J Acquir Immune Defic Syndr. 2013 May 1;63(1):77-85. doi: 10.1097/QAI.0b013e31828ace69. PMID 23412015
- [Background] Zolopa A, Sax PE, DeJesus E, Mills A, Cohen C, Wohl D, Gallant JE, Liu HC, Plummer A, White KL, Cheng AK, Rhee MS, Szwarcberg J; GS-US-236-0102 Study Team. A randomized double-blind comparison of coformulated elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate versus efavirenz/emtricitabine/tenofovir disoproxil fumarate for initial treatment of HIV-1 infection: analysis of week 96 results. J Acquir Immune Defic Syndr. 2013 May 1;63(1):96-100. doi: 10.1097/QAI.0b013e318289545c. PMID 23392460
- [Background] Eron JJ Jr, Rockstroh JK, Reynes J, Andrade-Villanueva J, Ramalho-Madruga JV, Bekker LG, Young B, Katlama C, Gatell-Artigas JM, Arribas JR, Nelson M, Campbell H, Zhao J, Rodgers AJ, Rizk ML, Wenning L, Miller MD, Hazuda D, DiNubile MJ, Leavitt R, Isaacs R, Robertson MN, Sklar P, Nguyen BY; QDMRK Investigators. Raltegravir once daily or twice daily in previously untreated patients with HIV-1: a randomised, active-controlled, phase 3 non-inferiority trial. Lancet Infect Dis. 2011 Dec;11(12):907-15. doi: 10.1016/S1473-3099(11)70196-7. Epub 2011 Sep 18. PMID 21933752
- [Background] German P, Warren D, West S, Hui J, Kearney BP. Pharmacokinetics and bioavailability of an integrase and novel pharmacoenhancer-containing single-tablet fixed-dose combination regimen for the treatment of HIV. J Acquir Immune Defic Syndr. 2010 Nov;55(3):323-9. doi: 10.1097/QAI.0b013e3181eb376b. PMID 20683270
- [Background] Zolopa AR, Berger DS, Lampiris H, Zhong L, Chuck SL, Enejosa JV, Kearney BP, Cheng AK. Activity of elvitegravir, a once-daily integrase inhibitor, against resistant HIV Type 1: results of a phase 2, randomized, controlled, dose-ranging clinical trial. J Infect Dis. 2010 Mar 15;201(6):814-22. doi: 10.1086/650698. PMID 20146631
- [Background] Schrijvers R, Debyser Z. Quad's in it for antiretroviral therapy? Lancet. 2012 Jun 30;379(9835):2403-2405. doi: 10.1016/S0140-6736(12)61029-0. No abstract available. PMID 22748575
- [Background] Cooper DA, Steigbigel RT, Gatell JM, Rockstroh JK, Katlama C, Yeni P, Lazzarin A, Clotet B, Kumar PN, Eron JE, Schechter M, Markowitz M, Loutfy MR, Lennox JL, Zhao J, Chen J, Ryan DM, Rhodes RR, Killar JA, Gilde LR, Strohmaier KM, Meibohm AR, Miller MD, Hazuda DJ, Nessly ML, DiNubile MJ, Isaacs RD, Teppler H, Nguyen BY; BENCHMRK Study Teams. Subgroup and resistance analyses of raltegravir for resistant HIV-1 infection. N Engl J Med. 2008 Jul 24;359(4):355-65. doi: 10.1056/NEJMoa0708978. PMID 18650513
- [Background] DeJesus E, Rockstroh JK, Henry K, Molina JM, Gathe J, Ramanathan S, Wei X, Yale K, Szwarcberg J, White K, Cheng AK, Kearney BP; GS-236-0103 Study Team. Co-formulated elvitegravir, cobicistat, emtricitabine, and tenofovir disoproxil fumarate versus ritonavir-boosted atazanavir plus co-formulated emtricitabine and tenofovir disoproxil fumarate for initial treatment of HIV-1 infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet. 2012 Jun 30;379(9835):2429-2438. doi: 10.1016/S0140-6736(12)60918-0. PMID 22748590
- [Background] Min S, Sloan L, DeJesus E, Hawkins T, McCurdy L, Song I, Stroder R, Chen S, Underwood M, Fujiwara T, Piscitelli S, Lalezari J. Antiviral activity, safety, and pharmacokinetics/pharmacodynamics of dolutegravir as 10-day monotherapy in HIV-1-infected adults. AIDS. 2011 Sep 10;25(14):1737-45. doi: 10.1097/QAD.0b013e32834a1dd9. PMID 21716073
- [Background] Min S, Song I, Borland J, Chen S, Lou Y, Fujiwara T, Piscitelli SC. Pharmacokinetics and safety of S/GSK1349572, a next-generation HIV integrase inhibitor, in healthy volunteers. Antimicrob Agents Chemother. 2010 Jan;54(1):254-8. doi: 10.1128/AAC.00842-09. Epub 2009 Nov 2. PMID 19884365
- [Background] Powderly WG. Integrase inhibitors in the treatment of HIV-1 infection. J Antimicrob Chemother. 2010 Dec;65(12):2485-8. doi: 10.1093/jac/dkq350. Epub 2010 Sep 18. PMID 20852268
- [Background] Song I, Borland J, Chen S, Patel P, Wajima T, Peppercorn A, Piscitelli SC. Effect of food on the pharmacokinetics of the integrase inhibitor dolutegravir. Antimicrob Agents Chemother. 2012 Mar;56(3):1627-9. doi: 10.1128/AAC.05739-11. Epub 2011 Dec 19. PMID 22183173
- [Background] Weller S, Chen S, Borland J, Savina P, Wynne B, Piscitelli SC. Bioequivalence of a dolutegravir, abacavir, and lamivudine fixed-dose combination tablet and the effect of food. J Acquir Immune Defic Syndr. 2014 Aug 1;66(4):393-8. doi: 10.1097/QAI.0000000000000193. PMID 24798770
- [Background] Raffi F, Jaeger H, Quiros-Roldan E, Albrecht H, Belonosova E, Gatell JM, Baril JG, Domingo P, Brennan C, Almond S, Min S; extended SPRING-2 Study Group. Once-daily dolutegravir versus twice-daily raltegravir in antiretroviral-naive adults with HIV-1 infection (SPRING-2 study): 96 week results from a randomised, double-blind, non-inferiority trial. Lancet Infect Dis. 2013 Nov;13(11):927-35. doi: 10.1016/S1473-3099(13)70257-3. Epub 2013 Sep 25. PMID 24074642
- [Background] Walmsley SL, Berenguer J, Kuong-Josses M-A, Kilby JM, Lutz T, Podzamczer D, et al. Dolutegravir Regimen Statistically Superior to Efavirenz/Tenofovir/Emtricitabine: 96-Week Results From the SINGLE Study (ING114467) In: 21st Conference on Retroviruses and Opportunistic Infections. Boston, MA; 2014.
- [Background] Cahn P, Pozniak AL, Mingrone H, Shuldyakov A, Brites C, Andrade-Villanueva JF, Richmond G, Buendia CB, Fourie J, Ramgopal M, Hagins D, Felizarta F, Madruga J, Reuter T, Newman T, Small CB, Lombaard J, Grinsztejn B, Dorey D, Underwood M, Griffith S, Min S; extended SAILING Study Team. Dolutegravir versus raltegravir in antiretroviral-experienced, integrase-inhibitor-naive adults with HIV: week 48 results from the randomised, double-blind, non-inferiority SAILING study. Lancet. 2013 Aug 24;382(9893):700-8. doi: 10.1016/S0140-6736(13)61221-0. Epub 2013 Jul 3. PMID 23830355
- [Background] Castagna A, Maggiolo F, Penco G, Wright D, Mills A, Grossberg R, Molina JM, Chas J, Durant J, Moreno S, Doroana M, Ait-Khaled M, Huang J, Min S, Song I, Vavro C, Nichols G, Yeo JM; VIKING-3 Study Group. Dolutegravir in antiretroviral-experienced patients with raltegravir- and/or elvitegravir-resistant HIV-1: 24-week results of the phase III VIKING-3 study. J Infect Dis. 2014 Aug 1;210(3):354-62. doi: 10.1093/infdis/jiu051. Epub 2014 Jan 19. PMID 24446523
- [Background] Clotet B, Feinberg J, van Lunzen J, Khuong-Josses MA, Antinori A, Dumitru I, Pokrovskiy V, Fehr J, Ortiz R, Saag M, Harris J, Brennan C, Fujiwara T, Min S; ING114915 Study Team. Once-daily dolutegravir versus darunavir plus ritonavir in antiretroviral-naive adults with HIV-1 infection (FLAMINGO): 48 week results from the randomised open-label phase 3b study. Lancet. 2014 Jun 28;383(9936):2222-31. doi: 10.1016/S0140-6736(14)60084-2. Epub 2014 Apr 1. PMID 24698485
- [Background] Walmsley SL, Antela A, Clumeck N, Duiculescu D, Eberhard A, Gutierrez F, Hocqueloux L, Maggiolo F, Sandkovsky U, Granier C, Pappa K, Wynne B, Min S, Nichols G; SINGLE Investigators. Dolutegravir plus abacavir-lamivudine for the treatment of HIV-1 infection. N Engl J Med. 2013 Nov 7;369(19):1807-18. doi: 10.1056/NEJMoa1215541. PMID 24195548
- [Background] Pilcher CD, Fiscus SA, Nguyen TQ, Foust E, Wolf L, Williams D, Ashby R, O'Dowd JO, McPherson JT, Stalzer B, Hightow L, Miller WC, Eron JJ Jr, Cohen MS, Leone PA. Detection of acute infections during HIV testing in North Carolina. N Engl J Med. 2005 May 5;352(18):1873-83. doi: 10.1056/NEJMoa042291. PMID 15872202
- [Background] D:A:D Study Group; Sabin CA, Worm SW, Weber R, Reiss P, El-Sadr W, Dabis F, De Wit S, Law M, D'Arminio Monforte A, Friis-Moller N, Kirk O, Pradier C, Weller I, Phillips AN, Lundgren JD. Use of nucleoside reverse transcriptase inhibitors and risk of myocardial infarction in HIV-infected patients enrolled in the D:A:D study: a multi-cohort collaboration. Lancet. 2008 Apr 26;371(9622):1417-26. doi: 10.1016/S0140-6736(08)60423-7. Epub 2008 Apr 2. PMID 18387667
- [Background] Costagliola D, Lang S, Mary-Krause M, Boccara F. Abacavir and cardiovascular risk: reviewing the evidence. Curr HIV/AIDS Rep. 2010 Aug;7(3):127-33. doi: 10.1007/s11904-010-0047-3. PMID 20521126
- See also: University of North Carolina website — http://www.unc.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- DTG/3TC/ABC FDC: Dolutegravir (DTG 50 mg), abacavir sulfate (ABC 600 mg) and lamivudine (3TC 300 mg) formulated in a single tablet fixed dose combination (FDC) (DTG/ABC/3TC, GSK2619619), administered orally, once daily initiated during acute HIV infection.
Period: Overall Study
Arm/Group | DTG/3TC/ABC FDC
Started | 40
Enrolled (Pending HLA and Hepatitis B results) | 40
Initiated Treatment | 37
Completed Week 24 | 34
Completed Week 48 | 33
Completed Week 96 (Two participants had data collected outside of Week 96 window) | 30
Completed | 30
Not Completed | 10
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | DTG/3TC/ABC FDC
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 26 [18 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37
Baseline CD4 Count [Median (Full Range); unit: cells/mm^3] | 478 [67 to 860]
Baseline HIV-1 RNA PCR Level [Median (Full Range); unit: copies/mL] | 382000 [1860 to 10000000]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Viral Load Measurement <200 Copies/mL at Week 24
Description: Total number of participants on study at Week 24 with an HIV-1 RNA level less than 200 copies/mL
Time Frame: Week 24
Population: Excludes 3 participants who terminated prior to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC/ABC FDC
Number analyzed (Participants) | 34
Participants | 34

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Event (AE)
Description: Sign/symptom, lab toxicity, or clinical events, or Grade 3 or higher AE that is definitely, probably, or possibly related to study treatment
Time Frame: Baseline through Week 96
Population: Two participants had data collected outside of Week 96 window
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC/ABC FDC
Number analyzed (Participants) | 37
Participants | 1

3. Secondary Outcome: Proportion of Treated Participants With HIV-1 RNA to <50 Copies/mL at Week 48
Description: Proportion of participants completing Week 48 with an HIV-1 RNA level less than 50 copies/mL
Time Frame: Week 48
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | DTG/3TC/ABC FDC
Number analyzed (Participants) | 33
proportion of participants | 0.88 [0.72 to 0.97]

4. Secondary Outcome: Median Change HIV-1 RNA Level Among Participants Completing Week 24 Visit
Time Frame: Baseline, Week 24
Population: Excludes 3 participants who terminated prior to Week 24
Measure: Median (Full Range); unit: copies/mL
Arm/Group | DTG/3TC/ABC FDC
Number analyzed (Participants) | 34
copies/mL | -590211 [-9999980 to -1830]

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent throughout treatment, a total of approximately 96 weeks.
Arm/Group | DTG/3TC/ABC FDC
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 5/37
Other Adverse Events (participants affected / at risk) | 21/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG/3TC/ABC FDC (N=37)
Exacerbation of Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Bronchitis (Infections and infestations) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Acute Stress Reaction (Psychiatric disorders) | 1 (1)
Chest Pain associated with Back Pain (General disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Anterior Uveitis (Eye disorders) | 1 (1)
Left Scrotal Cellulitis (Infections and infestations) | 1 (1)
Left Scrotal Abscess (Infections and infestations) | 1 (1)
Diabetic Ketoacidosis without coma associated with T1DM (Metabolism and nutrition disorders) | 1 (1)
Elevated Alanine Aminotransferase (ALT) (Investigations) | 1 (1)
Elevated Aspartate Aminotransferase (AST) (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG/3TC/ABC FDC (N=37)
ALT Increased (Investigations) | 3 (3)
Citrate Sensitivity (Injury, poisoning and procedural complications) | 2 (4)
Creatinine Clearance Decreased (Investigations) | 7 (8)
Headache (Nervous system disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (8)
Elevated BP During Leukapheresis (Injury, poisoning and procedural complications) | 13 (16)
IV Infiltration During Leukapheresis (General disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT02384395/Prot_SAP_000.pdf